CLINICAL TRIAL: NCT06331741
Title: Application of Collagen in Treatment of the Consequences of Injuries and Diseases of the Musculoskeletal System
Brief Title: Collagen for Treatment of Musculoskeletal Injuries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0403
Record Dates: First submitted 2024-03-07; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Anterior Cruciate Ligament Injuries; Hallux Rigidus
Keywords: anterior cruciate ligament; hallux rigidus; ACL reconstruction; collagen membrane; collagen matrix
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Hallux Rigidus | interventions — Anterior Cruciate Ligament Reconstruction; Control Groups

STUDY DESIGN:
Intervention Model Description: Main group for ACL: 5 patients with ACL injury, who undergo ACL reconstruction with collagen membrane augmentation; Reference group for ACL: 5 patients with ACL injury, who undergo ACL reconstruction without collagen membrane augmentation; Main group for HR (Hallux Rigidus): 5 patients with Hallux Rigidus, who undergo resection arthroplasty with introduction of collagen membrane Reference group: none
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The 1st group (Other): ACL reconstruction + collagen membrane
  Interventions: Procedure: Anterior cruciate ligament reconstruction, using graft, augmented with collagen membrane
- The 2nd group (Other): ACL reconstruction (control)
  Interventions: Procedure: Anterior cruciate ligament reconstruction, using graft, not augmented with collagen membrane (control group)
- The 3rd group (Other): Hallux Rigidus + collagen membrane
  Interventions: Procedure: Resection arthroplasty of the first metatarsophalangeal joint with the introduction of a collagen membrane into the joint cavity

INTERVENTIONS:
Procedure: Anterior cruciate ligament reconstruction, using graft, augmented with collagen membrane — Wrapping graft (tendon of the long fibular muscle) with collagen membrane before implantation
  Arms: The 1st group
Procedure: Anterior cruciate ligament reconstruction, using graft, not augmented with collagen membrane (control group) — Implantation of the native graft (tendon of the long fibular muscle) without any augmentation method
  Arms: The 2nd group
Procedure: Resection arthroplasty of the first metatarsophalangeal joint with the introduction of a collagen membrane into the joint cavity — Arthroplasty with consequent collagen membrane implantation
  Arms: The 3rd group

SUMMARY:
The purpose of the study:

Evaluation of the clinical efficacy and safety of the use of collagen matrix/membrane in the surgical treatment of the consequences of injuries and diseases of the musculoskeletal system (anterior cruciate ligament tears, rigid first toe) by using IKDC, KOOS, ACLOAS, VAS, AOFAS, SF-36 scales

DETAILED DESCRIPTION:
Application of Collagen in Treatment of the Consequences of Injuries and Diseases of the Musculoskeletal System

Indications:

* Damage to the anterior cruciate ligament (ACL) of the knee joint
* Rigid first toe

Research centers:

University Clinical Hospital No. 1 of the First Sechenov Moscow State Medical University (Sechenov University)

The product under study:

The collagen membrane

Specifications:

-The product is a membrane made of type 1 collagen obtained from the ligaments of cattle. Chemically cross-linked with glutaraldehyde. The size of the membrane is 15x4x0.3 cm in dry form (can be adjusted depending on the patient's need).

Product shape: tape (medical device) Composition: type 1 collagen Packaging: in a sterilization bag Transportation: in a dry place, protected from light, at a temperature of 10 to 30 °C.

Shelf life: 2 years Storage: in a dry place, protected from light, at a temperature of 10 to 30 °C. Purpose: for implantation Storage conditions of the product: in a dry place, protected from light, at a temperature from 10 to 30 °C. Soak in saline solution for 10 minutes before use.

Sterilization: Steripak electron beam sterilization Manufacturer: Sechenov First Moscow State Medical University of the Ministry of Health of the Russian Federation (Sechenov University)

Research objectives:

Tasks for the reconstruction of the ACL using a collagen membrane:

1. Change in the score of the Form for registering the results of the knee joint examination of the International Knee Documentation Committee (IKDC);
2. Change in the score of the Knee injury and Osteoarthritis Outcome Score (KOOS) relative to the baseline level;
3. Change in the score of the Modified Lysholm scale relative to the initial level;
4. Assessment of the condition of the transplant based on the results of control MRI data, measured on Anterior Cruciate Ligament OsteoArthritis Score (ACLOAS)

Tasks for the application of collagen spacer of the first metatarsophalangeal joint:

1. Formation of clinical groups of patients with 3-4 stages of Hallux rigidus.
2. The development of personalized collagen, the formation of a membrane of the required size
3. Formation of a unified protocol of the operational manual
4. Development of a program of postoperative orthopedic regimen and rehabilitation

Assessment of the formation of syndesmosis by using instrumental research methods

Safety assessment parameters:

The frequency of adverse events and serious adverse events according to subjective complaints, physical examination, vital signs, ECG (Electrocardiography) and laboratory tests against the background of treatment using the technique of collagen membrane transplantation

The study population:

For the reconstruction of the anterior cruciate ligament using a collagen membrane:

men and women from 18 to 60 years old, with partial or complete damage to the anterior cruciate ligament, who will undergo autograft surgery, will be included in the work

For the collagen spacer of the first toe:

men and women from 18 to 60 years old, with 3-4 stages of Hallux rigidus, who will undergo resection arthroplasty with the introduction of a biocompatible collagen spacer into the joint cavity, will be included in the work

Number of patients:

10 patients with ACL damage 5 patients with a rigid first toe

Duration of the study:

For each patient - 12 months.

Research methodology:

Design for the reconstruction of the ACL using a collagen membrane:

The design involves the study of the medical device in experimental treatment groups in comparison with the control group.

The study group will initially include 5 patients. As a reference group, the results of treatment of 5 patients with ACL reconstruction by autograft.

Design for the collagen spacer of the first toe:

The study group will initially include 5 patients.

Description of the work stages:

For ACL reconstruction using a collagen membrane:

Screening:

* Procedure for obtaining informed consent;
* Collection of demographic data, medical history; registration of previous surgical interventions on the knee joint;
* Assessment of vital signs (blood pressure, heart rate, respiratory rate, t°);
* Measurement of height, body weight, body mass index (BMI) (growth is estimated once per study - at screening);
* Physical examination;
* Evaluation of MRI of the knee joint (ACLOAS);
* Registration of the previous/concomitant therapy;
* Registration of pain therapy;
* Assessment of compliance with the inclusion/non-inclusion criteria;

For patients who meet the preliminary inclusion criteria and do not meet any of the criteria for non-inclusion in the screening, the date and time of arthroscopy will be assigned.

The researcher gives the patient:

* Patient information sheet and informed consent form;
* Patient's card;
* Rehabilitation program.

Hospitalization:

Day 1

* Assessment of vital signs (blood pressure, heart rate, respiratory rate, t°);
* Measurement of body weight, BMI;
* Physical examination;
* Patients will be assessed according to the following scales: the Knee injury and Osteoarthritis Outcome Score (KOOS), the International Knee Documentation Committee (IKDC), assessment on the Modified Lysholm Scale
* Assessment of compliance with the inclusion/non-inclusion criteria;
* Assessment of exclusion criteria;

Day 2 Surgical treatment: ligament reconstruction. After surgery, adverse events, concomitant therapy, pain therapy, and vital signs will be re-evaluated.

Day 3-7 (Discharge)

* Assessment of adverse events, exclusion criteria, concomitant therapy, pain therapy;
* assessment of vital signs (blood pressure, heart rate, respiratory rate, t°);
* Providing instructions on the prescribed rehabilitation program;
* discharge from the hospital.

Observation period Visit 1 (Week 2)

* Removal of postoperative sutures
* Assessment of the implementation of the prescribed rehabilitation program;
* Providing further instructions on the prescribed rehabilitation program;
* Assessment of vital signs (blood pressure, heart rate, respiratory rate, t°);
* Measurement of body weight, BMI;
* Physical examination;

Visit 2 (Week 6)

* Assessment of the implementation of the prescribed rehabilitation program;
* Providing further instructions on the rehabilitation program;
* Assessment of vital signs (blood pressure, heart rate, respiratory rate, t°);
* Physical examination;
* Assessment according to the following scales: the Knee injury and Osteoarthritis Outcome Score (KOOS), the International Knee Documentation Committee (IKDC)
* Assessment on the Modified Lysholm scale;
* MRI of the operated knee joint (ACLOAS);
* Preparation of an interim report to assess the safety of the material (for the first patient included in the study).

Visit 3 (Week 24-48)

* Assessment of the implementation of the prescribed rehabilitation program;
* Providing instructions on the prescribed rehabilitation program;
* Assessment of vital signs (blood pressure, heart rate, respiratory rate, t°);
* Measurement of body weight, BMI;
* Physical examination;
* Assessment according to the following scales: the Knee injury and Osteoarthritis Outcome Score (KOOS), the International Knee Documentation Committee (IKDC)
* Assessment on the Modified Lysholm scale;
* MRI of the operated knee joint (ACLOAS).

For the collagen spacer of the first toe

Screening:

* Procedure for obtaining informed consent;
* Collection of demographic data, medical history;
* Assessment of vital signs (blood pressure, heart rate, respiratory rate, t°);
* Measurement of height, body weight, body mass index (BMI) (growth is estimated once per study - at screening);
* Physical examination;
* Evaluation of foot radiographs in two projections, functional MSCT (Multislice spiral computed tomography) of the foot
* Registration of the previous/concomitant therapy;
* Registration of pain therapy;
* Assessment of compliance with the inclusion/non-inclusion criteria;

For patients who meet the preliminary inclusion criteria and do not meet any of the criteria for non-inclusion in the screening, the date and time of the operation will be assigned.

The researcher gives the patient:

* Patient information sheet and informed consent form;
* Patient's card;

Hospitalization:

Day 1

* Assessment of vital signs (blood pressure, heart rate, respiratory rate, t°);
* Measurement of body weight, BMI;
* Physical examination;
* Patients will be evaluated according to the scales: VAS (visual analog pain scale), AOFAS (American Orthopaedic Foot and Ankle Society, Ankle-Hindfoot Score), SF-36 (36-Item Short Form Survey)
* Assessment of compliance with the inclusion/non-inclusion criteria;
* Assessment of exclusion criteria

Day 2 Surgical treatment: resection arthroplasty of the first metatarsophalangeal joint with implantation of a collagen spacer. After the operation, adverse events will be re-evaluated, symptomatic, analgesic therapy will be performed, and vital signs will be dynamically evaluated.

* Dressing of the postoperative wound
* Performing a control radiography of the operated feet in two projections
* Learning to walk in orthopedic shoes

Day 3-7 (Discharge)

* Assessment of adverse events, symptomatic, analgesic therapy;
* assessment of vital signs (blood pressure, heart rate, respiratory rate, t°);
* Walking in orthopedic shoes under the supervision of the attending physician;
* Dressing of the postoperative wound
* discharge from the hospital.

The observation period.

1. Visit 1 (Week 2)

   * Clinical examination
   * Filling in evaluation scales by the patient
   * Dressing of the postoperative wound, removal of stitches
   * Performing a control radiography of the operated feet in two projections
   * Evaluation of results (data from evaluation scales (VAS, AOFAS, SF-36), evaluation of functional and radiological results)
2. Visit 2 (Week 4)

   * Clinical examination
   * Filling in evaluation scales by the patient
   * Performing a control radiography of the operated feet in two projections
   * Evaluation of the results (data from evaluation scales (VAS, AOFAS, SF-36), assessment of pain syndrome and amplitude of back flexion in the metatarsophalangeal joint and radiological result)
3. Visit 3 (Week 8)

   * Clinical examination
   * Filling in evaluation scales by the patient
   * Performing a control radiography of the operated feet in two projections
   * Evaluation of the results (data from evaluation scales (VAS, AOFAS, SF-36), assessment of pain syndrome and amplitude of back flexion in the metatarsophalangeal joint and radiological result)

ELIGIBILITY:
Inclusion criteria:

For ACL reconstruction groups:

* Type of damage (rupture of the anterior cruciate ligament (complete or partial);
* Availability of an informed consent form signed and dated by the patient.
* The patient's understanding of the strict requirements of the protocol, rehabilitation program and follow-up program and the desire to follow them.
* The patient's consent to the use of the following drugs: nonsteroidal anti-inflammatory drugs (NSAIDs) (according to indications); antibiotics; anticoagulants.

For collagen membrane of the first toe:

* The type of degenerative disease of the first metatarsophalangeal joint is Hallux rigidus of stage 3-4.
* Availability of an informed consent form signed and dated by the patient.
* The patient's understanding of the strict requirements of the protocol, rehabilitation program and follow-up program and the desire to follow them.
* The patient's consent to the use of the following drugs: nonsteroidal anti-inflammatory drugs (NSAIDs) (according to indications); antibiotics; anticoagulants

Non-inclusion criteria:

* Abuse of alcohol or narcotic substances (medicines).
* Any clinically significant or symptomatic vascular or neurological disease of the lower extremities.
* The presence of rheumatoid arthritis, parainfectious or infectious arthritis and the condition after the listed diseases, as well as the following diseases in the area of the damaged knee joint: septic arthritis, inflammatory joint disease, recurrent pseudopodagra, Paget's disease, ochronosis, acromegaly, hemochromatosis, Wilson-Konovalov disease, primary osteochondromatosis, hereditary diseases, mutation of collagen genes.
* Pregnancy and planned pregnancy (inability to perform MRI), lactation period.
* Obesity (body mass index > 30 kg/m2).
* Uncontrolled diabetes mellitus.
* Significant cardiovascular diseases currently or within 12 months prior to screening, including: chronic heart failure of class III or IV (according to the classification of the New York Cardiological Association), severe arrhythmia requiring treatment with antiarrhythmic drugs of classes Ia, Ib, Ic or III, unstable angina pectoris, myocardial infarction, heart and coronary surgery blood vessels, significant diseases of the heart valves, uncontrolled arterial hypertension with systolic blood pressure > 180 mmHg and diastolic blood pressure > 110 mmHg, pulmonary embolism or deep vein thrombosis;
* Significant thyroid dysfunction in the decompensation stage;
* Any uncontrolled concomitant somatic disease, including through a stable therapy regimen;
* Nephrotic syndrome, moderate to severe chronic renal failure, or significant kidney disease with creatinine levels > 1.5 mg/dl (132 mmol/l) in men and > 1.4 mg/dl (123 mmol/l) in women or glomerular filtration rate (GFR) < 60 ml/min;
* Current diagnosis of osteomyelitis and (or) infection with human immunodeficiency virus (HIV-1, HIV-2) and (or) hepatitis C virus (HCV) and (or) hepatitis B virus (HBV) and (or) syphilis. An increase in AST (aspartate transaminase), ALT (alanine transaminase) or alkaline phosphatase of serum ≥ 2.5 times from the upper limit of the norm; an increase in the level of total bilirubin ≥ 2 times from the upper limit of the norm;

Exclusion criteria:

* The patient's refusal to participate in the study;
* The development of an allergic reaction to the product;
* Loss of contact with the patient for further observation;
* The decision of the research physician to terminate the patient's participation in the study prematurely if, in the opinion of the researcher, the patient cannot continue further participation in the study for any reason.
* Inclusion in the study in violation of the inclusion/non-inclusion criteria.
* Significant protocol violations that may affect patient safety and/or the integrity of the study data (in consultation with the medical monitor).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
The International Knee Documentation Committee score | 1,5 and 6 months postoperatively
  Change in the score of the Form for registering the results of the knee joint examination of the The International Knee Documentation Committee (IKDC) for ACL groups values: min - 0 points (0%); max - 87 points (100%) The higher score means better outcome
The Knee injury and Osteoarthritis Outcome Score | 1,5 and 6 months postoperatively
  Change in the score of the Knee injury and Osteoarthritis Outcome Score (KOOS) for ACL groups values: min - 0%; max - 100% The higher score means better outcome
Modified Lysholm scale | 1,5 and 12 months postoperatively
  Change in the score of the Modified Lysholm scale for ACL groups values: min - 0%; max - 100% The higher score means better outcome
Anterior Cruciate Ligament OsteoArthritis Score | 6 months postoperatively
  Assessment of the condition of the transplant based on the results of control MRI data measured on Anterior Cruciate Ligament OsteoArthritis Score (ACLOAS) for ACL groups values: min - 0 points; max - 3 points The higher score means worse outcome
American Orthopaedic Foot and Ankle Society, Ankle-Hindfoot Score | 2, 4 and 8 weeks postoperatively
  American Orthopaedic Foot and Ankle Society, Ankle-Hindfoot Score (AOFAS) for Hallux Rigidus group values: min - 0 points (0%); max - 100 points (100%) The higher score means better outcome
36-Item Short Form Survey | 2, 4 and 8 weeks postoperatively
  36-Item Short Form Survey (SF-36) for Hallux Rigidus group values: min - (0%); max - (100%) The higher score means better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Alexey V Lychagin, MD, PhD, Study Chair — IM Sechenov University
Locations (1):
- university clinical hospital № 1I.M.Sechenov First Moscow State Medical University. The Department of Traumatology, Orthopedics and Disaster Surgery, Moscow, Russia